CLINICAL TRIAL: NCT01332565
Title: An Open-Label, Single Dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of GSK1349572 (Dolutegravir, DTG) in Healthy Japanese Subjects
Brief Title: A Study to Investigate the Pharmacokinetics, Safety and Tolerability of GSK1349572 (Dolutegravir, DTG) in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 115381
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1349572; pharmacokinetics; Japanese; HIV
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All subjects will receive a 50 mg single dose of GSK1349572
  Interventions: Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572 — 50mg tablet

SUMMARY:
This study is a Phase 1, open label, non-randomized, single dose study to determine pharmacokinetics, safety and tolerability of doultegravir (DTG) following 50 mg single oral administration in healthy Japanese subjects. A total of 10 healthy Japanese subjects will be enrolled in this study to receive a 50 mg single dose of DTG. Subjects will have a screening visit within 30 days prior to the administration of study drug, a treatment visit, and a follow-up visit 7-14 days after the administration of study drug.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* The subject is a healthy Japanese Japanese subjects who were born in Japan with 4 ethnic Japanese grandparents and must not have lived outside Japan for more than 5 years with being a Japanese passport holder. Healthy as judged by a responsible physician with no clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* The subject is greater than or equal to 20 and less than or equal to 55 years of age, inclusive.
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mIU/mL and estradiol < 40 pg/mL (< 147 pmol/L) is confirmatory]. Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for the time period between screening and dosing of study drugs to sufficiently minimize the risk of pregnancy at that point. Female subjects must also agree to use contraception throughout the study and until two weeks after the last dose of study medications.
* Body weight less than or equal to 50 kg (110 lbs.) for men and less than or equal to 45 kg (99 lbs.) for women and body mass index (BMI) between 18.5 to 28 kg/m2 inclusive.
* A signed and dated written informed consent is obtained from the subject prior to screening.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject's systolic blood pressure is outside the range of 90-140 mmHg, or diastolic blood pressure is outside the range of 45-90 mmHg or heart rate is outside the range of 45-100 bpm for both male and female subjects. The subject's body temperature is > 37.5 degrees celcius.
* History/evidence of symptomatic or asymptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or congenital cardiac diseases or any clinically significant cardiac diseases.
* An episode of cardiac syncope within one year before screening period.
* History/evidence of clinically significant pulmonary diseases and hyper/hypo-thyroidism.
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV-1 antibody result.
* Has a history of regular alcohol consumption averaging > 7 drinks/week for women or >14 drinks/week for men (1 drink (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of the screening visit.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample.
* Has a history of use of tobacco- or nicotine-containing products within 6 months of the screening visit.
* The subject has a positive pre-study drug and/or alcohol screen.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* History or presence of allergy or intolerance to the study drug or its components or drugs of its class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin induced thrombocytopenia should not be enrolled.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort and iron supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, or serum creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and pancreatitis should be excluded.
* History of significant renal or hepatic diseases.
* History of Gilbert's syndrome.
* Has an abnormal ECG as described in the protocol.
* Clinically significant anomaly in electrolytes in subjects with heart rate greater than or equal to 60/min

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma DTG pharmacokinetic parameters following single dose administration: area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC(0-t)). | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: area under the plasma concentration-time curve from time zero to infinity (AUC(0-∞)). | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: maximum observed concentration (Cmax). | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: concentration at 24h post-dose (C24). | for 72 hours

SECONDARY OUTCOMES:
Plasma DTG pharmacokinetic parameters following single dose administration: time to maximum observed concentration (tmax) | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: last quantifiable concentration (Ct). | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: terminal phase half-life (t½) | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: absorption lag time (tlag) | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: apparent clearance (CL/F) | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: mean residence time (MRT). | for 72 hours
Plasma DTG pharmacokinetic parameters following single dose administration: apparent volume of distribution (Vz/F). | for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Cypress, California, United States